CLINICAL TRIAL: NCT06486870
Title: Comparative Study Between Two Ovulation Induction Therapies and Laparoscopic Ovarian Drilling on Clinical Outcomes in Clomiphene Citrate-Resistant PCOS Women
Brief Title: Comparison Between Two Ovulation Induction Therapies and LOD on Clinical Outcomes in CC-Resistant PCOS Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA-2024-2
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
Keywords: gonadotropin; letrozole; clomiphene citrate; ovarian drilling; pregnancy rate; ovulation rate
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Gonadotropins; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- gonadotropin (Experimental): Human menopausal gonadotrophin (hMG) is given starting on cycle day three in a dose of 75 IU alternate days. The aim of treatment is to achieve mono-ovulation. Monitoring of treatment is achieved by serial transvaginal ultrasound scanning every other day starting from cycle day nine. Size and number of follicles is recorded in patients follow up sheets. The dose of hMG is reviewed around stimulation day 10 and if follicular development is unsatisfactory, the dose is increased to 75 IU daily .If a good response is not achieved day16 ; the cycle is cancelled. A new cycle is commenced with a higher starting dose of hMG (75 IU per day). When one follicle reached a size of > =18 mm a single dose of 10,000 IU human chorionic gonadotrophin (hCG, Pregnyl, Epifasi, Choriomon) is given.
  Interventions: Drug: Gonadotropin
- letrozole (Experimental): : 5 mg LE oral tablets are administered on the fifth day of menses and then every day for 5 days. Treatment is repeated for up to six cycles
  Interventions: Drug: Letrozole
- unilateral laparoscopic ovarian drilling (Experimental): Laparoscopic ovarian drilling will be done according to the following:
  Electrocautery using a mixed current in monopolar electrosurgical needle will be into introduced through the ovarian ipsilateral parts and applied up to 4 point cauterisation of the ovarian capsule, each for 4 second, at 40 W and for a diameter of 3mm and a depth of 4 mm in the antimesentric surface . (Amer et al 2003, Sawant S et al 2019) ,the procedure will be applied for one ovary .
  The patient under the study will be followed up to six months of continuous marital life after the procedure
  Interventions: Procedure: laparoscopic ovarian drilling

INTERVENTIONS:
Drug: Gonadotropin — Human menopausal gonadotrophin (hMG) is given starting on cycle day three in a dose of 75 IU alternate days. The aim of treatment is to achieve mono-ovulation. Monitoring of treatment is achieved by serial transvaginal ultrasound scanning every other day starting from cycle day nine. Size and number of follicles is recorded in patients follow up sheets. The dose of hMG is reviewed around stimulation day 10 and if follicular development is unsatisfactory, the dose is increased to 75 IU daily .If a good response is not achieved day16 ; the cycle is cancelled. A new cycle is commenced with a higher starting dose of hMG (75 IU per day). When one follicle reached a size of > =18 mm a single dose of 10,000 IU human chorionic gonadotrophin (hCG, Pregnyl, Epifasi, Choriomon) is given.
  Arms: gonadotropin
Drug: Letrozole — 5 mg LE oral tablets are administered on the fifth day of menses and then every day for 5 days. Treatment is repeated for up to six cycles
  Arms: letrozole
Procedure: laparoscopic ovarian drilling — Laparoscopic ovarian drilling will be done according to the following:
  Electrocautery using a mixed current in monopolar electrosurgical needle will be into introduced through the ovarian ipsilateral parts and applied up to 4 point cauterisation of the ovarian capsule, each for 4 second, at 40 W and for a diameter of 3mm and a depth of 4 mm in the antimesentric surface . (Amer et al 2003, Sawant S et al 2019) ,the procedure will be applied for one ovary .
  The patient under the study will be followed up to six months of continuous marital life after the procedure
  Arms: unilateral laparoscopic ovarian drilling

SUMMARY:
Polycystic ovary syndrome (PCOS) is a prevalent endocrine disorder affecting 4-8% of reproductive-aged women and is a leading cause of infertility due to oligo-anovulation (1). Studies suggest a higher prevalence of 17.8-19.9% based on Rotterdam diagnostic criteria. PCOS is diagnosed by the presence of at least two out of three criteria: oligo- and/or anovulation, hyperandrogenism, and polycystic ovaries, with other etiologies excluded (2). Clomiphene citrate (CC), a selective estrogen receptor modulator, has been the first-line treatment for inducing ovulation in anovulatory women with PCOS for decades. Approximately 80% of women resume ovulation with CC, but only 35-40% achieve pregnancy. About 15-40% of women are resistant to CC, defined as failure to ovulate after receiving a maximum dosage of 150 mg per day for 5 days starting on the third day of the menstrual cycle. For CC-resistant women, metformin, an insulin sensitizer, has been explored but shows limited effectiveness except in combination with CC. Gonadotropins are the standard treatment for CC-resistant PCOS but come with risks of multiple pregnancies and ovarian hyperstimulation syndrome (OHSS) (3). Letrozole, an aromatase inhibitor, is another treatment option that prevents the conversion of androgens to estrogen, thereby increasing gonadotropin-releasing hormone (GnRH) secretion and promoting ovulation. Letrozole has shown superior ovulation and live birth rates compared to CC and is now recommended as the first-line treatment for anovulation in women with PCOS. It has comparable rates of OHSS and miscarriage to CC, but fewer relevant studies have compared it directly to laparoscopic ovarian drilling (LOD) (4). LOD is an alternative to gonadotropins for inducing ovulation in CC-resistant PCOS. It involves surgical intervention, which can be either unilateral or bilateral, and is effective without the risks of multiple pregnancies or OHSS. LOD also increases ovarian responsiveness to CC. Despite minimal morbidity, LOD can lead to tubo-ovarian adhesions and premature ovarian failure, although these risks are reduced by careful technique (5).

DETAILED DESCRIPTION:
### Materials and Methods

**Design:** A randomized clinical study to evaluate and compare the effects of gonadotropins, Letrozole, and unilateral laparoscopic ovarian drilling in infertile women with PCOS. Conducted at Kasr El Aini Maternity Hospital, Cairo University, gynecological and infertility clinics.

**Patients:** The study includes infertile women aged 20-35 years with PCOS referred to the gynecology and infertility clinics of the Department of Obstetrics and Gynecology, Kasr Ainy Hospital, Cairo University. Women diagnosed with PCOS based on the Rotterdam criteria (ovulatory disturbance, hyperandrogenism, and the presence of more than 12 follicles, 2-9 mm in diameter, in each ovary by ultrasound examination) are randomly assigned to one of three groups: Letrozole (G1), Gonadotropin (G2), or Laparoscopic Unilateral Ovarian Drilling (G3), based on a computer-generated random number sequence. Side effects for each intervention are registered.

**Treatment Protocol:**

* Group I (G1): Letrozole 2.5 mg oral tablets, administered from the fifth day of menses for 5 days, repeated for up to six cycles.
* Group II (G2): Human menopausal gonadotropin (hMG) starts on cycle day three, 75 IU every other day, aiming for mono-ovulation. Monitoring through transvaginal ultrasound begins on cycle day nine. The hMG dose is adjusted based on follicular response. Cycles are cancelled for under or over-response.
* Group III (G3): Laparoscopic ovarian drilling with electrocautery (mixed current, monopolar electrosurgical needle, 4-point cauterization, each for 4 seconds, 40 W, 3 mm diameter, 4 mm depth) on one ovary.

**Follow-Up:** Patients will be monitored for six months post-intervention. Hormonal profiles will be reassessed at the end of the study period. Statistical analyses will be performed using Microsoft Excel 2007 and IBM SPSS version 22. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 35 years
* Infertile woman diagnosed to have PCO according to Rotterdam criteria as ovulatory distrbance, hyperandrogenism and presence of more than 12 follicles, 2- 9 mm in diameter in each other by ultrasound examination
* Resistance to clomiphene citrate i.e failed to respond to clomiphene citrate dose up to 150 mg per day for at least 3 cycles
* BMI from18-30
* High LH/FSH ratio≥1.5 , LH level ≥10IU/l)

Exclusion Criteria:

* Extremes of age less than 20 years old or more than 35 years old
* Hormonal therapy and oral contraception for the past 3cycle
* Other causes of infertility including tubal , uterine and male causes .
* Pre-existing endocrine disease including thyroid disorder, cushing's syndrome and congenital adrenal hyperplasia
* Any previous version surgery
* Obese patients with BMI >35
* Low ovarian reserve by AMH serum level measurement (AMH < .5-1.1 ng/ml).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — infertile women from 20 to 35 years old with PCOS referred to gynecology and infertility clinics, Department of Obstetrics and Gynecology,Kasr Ainy Hospital , Cairo University. Infertile woman diagnosed to have PCO according to Rotterdam criteria as ovulatory disturbance, hyperandrogenism and presence of more than 12 follicles, 2- 9 mm in diameter in each other by ultrasound examination
Enrollment: 183 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 6 month
  identified by serum β-HCG of >50 IU/L and gestational sac seen on ultrasound.

SECONDARY OUTCOMES:
ovulation rate | 6 months
  The ovulation rate refers to the percentage of women who successfully ovulate after a particular treatment regimen during a specified time period.
multiple pregnancy rate | 6 months
  The multiple pregnancy rate refers to the percentage of pregnancies that result in the birth of more than one baby, such as twins, triplets, or higher-order multiples, following a particular fertility treatment.
miscarriage rate | 6 months
  The miscarriage rate refers to the percentage of pregnancies that end in miscarriage, defined as the spontaneous loss of a pregnancy before the fetus reaches viability (usually before 20 weeks of gestation).

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh Sheeba, MD, Study Director — kasr alainy, Cairo university
Locations (1):
- faculty of medicine, Kasr el ainy hospital, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomas S, Woo I, Ho J, Jones T, Paulson R, Chung K, Bendikson K. Ovulation rates in a stair-step protocol with Letrozole vs clomiphene citrate in patients with polycystic ovarian syndrome. Contracept Reprod Med. 2019 Dec 9;4:20. doi: 10.1186/s40834-019-0102-4. eCollection 2019. PMID 31867117
- [Result] Yildiz BO, Bozdag G, Yapici Z, Esinler I, Yarali H. Prevalence, phenotype and cardiometabolic risk of polycystic ovary syndrome under different diagnostic criteria. Hum Reprod. 2012 Oct;27(10):3067-73. doi: 10.1093/humrep/des232. Epub 2012 Jul 9. PMID 22777527
- [Result] Brown J, Farquhar C. Clomiphene and other antioestrogens for ovulation induction in polycystic ovarian syndrome. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD002249. doi: 10.1002/14651858.CD002249.pub5. PMID 27976369
- [Result] Yang AM, Cui N, Sun YF, Hao GM. Letrozole for Female Infertility. Front Endocrinol (Lausanne). 2021 Jun 16;12:676133. doi: 10.3389/fendo.2021.676133. eCollection 2021. PMID 34220713
- [Result] Liu W, Dong S, Li Y, Shi L, Zhou W, Liu Y, Liu J, Ji Y. Randomized controlled trial comparing letrozole with laparoscopic ovarian drilling in women with clomiphene citrate-resistant polycystic ovary syndrome. Exp Ther Med. 2015 Oct;10(4):1297-1302. doi: 10.3892/etm.2015.2690. Epub 2015 Aug 19. PMID 26622481
- [Result] Moazami Goudarzi Z, Fallahzadeh H, Aflatoonian A, Mirzaei M. Laparoscopic ovarian electrocautery versus gonadotropin therapy in infertile women with clomiphene citrate-resistant polycystic ovary syndrome: A systematic review and meta-analysis. Iran J Reprod Med. 2014 Aug;12(8):531-8. PMID 25408702
- [Result] Davar R, Tabibnejad N, Kalantar SM, Sheikhha MH. The luteinizing hormone beta-subunit exon 3 (Gly102Ser) gene mutation and ovarian responses to controlled ovarian hyperstimulation. Iran J Reprod Med. 2014 Oct;12(10):667-72. PMID 25469124
- [Result] Thessaloniki ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Consensus on infertility treatment related to polycystic ovary syndrome. Hum Reprod. 2008 Mar;23(3):462-77. doi: 10.1093/humrep/dem426. PMID 18308833
- [Result] Godinjak Z, Javoric R. Clinical outcome and hormone profiles before and after laparoscopic electroincision of the ovaries in women with polycystic ovary syndrome. Bosn J Basic Med Sci. 2007 May;7(2):171-5. doi: 10.17305/bjbms.2007.3076. PMID 17489756
- [Result] Abu Hashim H, Al-Inany H, De Vos M, Tournaye H. Three decades after Gjonnaess's laparoscopic ovarian drilling for treatment of PCOS; what do we know? An evidence-based approach. Arch Gynecol Obstet. 2013 Aug;288(2):409-22. doi: 10.1007/s00404-013-2808-x. Epub 2013 Mar 30. PMID 23543241
- [Result] Ibrahim MH, Tawfic M, Hassan MM, Sedky OH. Letrozole versus laparoscopic ovarian drilling in infertile women with PCOS resistant to clomiphene citrate. Middle East Fertility Society Journal. 2017 Dec 1;22(4):251-4.
- [Result] Abdellah MS. Reproductive outcome after letrozole versus laparoscopic ovarian drilling for clomiphene-resistant polycystic ovary syndrome. Int J Gynaecol Obstet. 2011 Jun;113(3):218-21. doi: 10.1016/j.ijgo.2010.11.026. Epub 2011 Apr 1. PMID 21457973
- [Result] Elnashar A, Abdelmageed E, Fayed M, Sharaf M. Clomiphene citrate and dexamethazone in treatment of clomiphene citrate-resistant polycystic ovary syndrome: a prospective placebo-controlled study. Hum Reprod. 2006 Jul;21(7):1805-8. doi: 10.1093/humrep/del053. Epub 2006 Mar 16. PMID 16543255
- [Result] Yadav P, Singh S, Singh R, Jain M, Awasthi S, Raj P. To study the effect on fertility outcome by gonadotropins vs laparoscopic ovarian drilling in clomiphene-resistant cases of polycystic ovarian syndrome. Journal of the South Asian Federation of Obstetrics and Gynaecology. 2017 Oct;9(4):336-40.
- [Result] Mehrabian F, Eessaei F. The laparoscopic ovarian electrocautery versus gonadotropin therapy in infertile women with clomiphene citrate-resistant polycystic ovary syndrome; a randomized controlled trial. J Pak Med Assoc. 2012 Mar;62(3 Suppl 2):S42-4. PMID 22768457
- [Result] Ganesh A, Goswami SK, Chattopadhyay R, Chaudhury K, Chakravarty B. Comparison of letrozole with continuous gonadotropins and clomiphene-gonadotropin combination for ovulation induction in 1387 PCOS women after clomiphene citrate failure: a randomized prospective clinical trial. J Assist Reprod Genet. 2009 Jan;26(1):19-24. doi: 10.1007/s10815-008-9284-4. Epub 2009 Jan 7. PMID 19127427